CLINICAL TRIAL: NCT01777152
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study of Brentuximab Vedotin and CHP (A+CHP) Versus CHOP in the Frontline Treatment of Patients With CD30-positive Mature T-cell Lymphomas
Brief Title: ECHELON-2: A Comparison of Brentuximab Vedotin and CHP With Standard-of-care CHOP in the Treatment of Patients With CD30-positive Mature T-cell Lymphomas
Acronym: ECHELON-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGN35-014; 2012-002751-42 (EudraCT Number)
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Anaplastic Large-Cell Lymphoma; Non-Hodgkin Lymphoma; T-Cell Lymphoma
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Drug Therapy; Hematologic Diseases; Lymphoma; Monomethyl auristatin E; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Doxorubicin; Prednisone; Vincristine; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHOP (Active Comparator): cyclophosphamide, doxorubicin, vincristine, and prednisone
  Interventions: Drug: doxorubicin; Drug: prednisone; Drug: vincristine; Drug: cyclophosphamide
- A+CHP (Experimental): brentuximab vedotin, cyclophosphamide, doxorubicin, and prednisone
  Interventions: Drug: brentuximab vedotin; Drug: doxorubicin; Drug: prednisone; Drug: cyclophosphamide

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg every 3 weeks by IV infusion for 6-8 cycles
  Other Names: Adcetris; SGN-35
  Arms: A+CHP
Drug: doxorubicin — 50 mg/m2 every 3 weeks by IV infusion for 6-8 cycles
Drug: prednisone — 100 mg on Days 1 to 5 of each 3-week cycle, orally for 6-8 cycles
Drug: vincristine — 1.4 mg/m2 (maximum 2 mg) every 3 weeks by IV infusion for 6-8 cycles
  Arms: CHOP
Drug: cyclophosphamide — 750 mg/m2 every 3 weeks by IV infusion for 6-8 cycles

SUMMARY:
This is a double-blind, randomized, multicenter, phase 3 clinical trial to compare the efficacy and safety of brentuximab vedotin in combination with CHP with the standard-of-care CHOP in patients with CD30-positive mature T-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, CD30-positive mature T-cell lymphomas
* Fluorodeoxyglucose (FDG)-avid disease by PET and measurable disease of at least 1.5 cm by CT
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

Exclusion Criteria:

* History of another primary invasive malignancy that has not been in remission for at least 3 years
* Current diagnosis of primary cutaneous CD30-positive T-cell lymphoproliferative disorders and lymphomas or mycosis fungoides
* History of progressive multifocal leukoencephalopathy (PML)
* Cerebral/meningeal disease related to the underlying malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Manley, MD, Study Director — Seagen Inc.
Locations (144):
- United States (32):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Shands Cancer Center / University of Florida, Gainesville, Florida
  - Orlando Health, Inc., Orlando, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Holden Comprehensive Cancer Center / University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - James P. Wilmot Cancer Center / University of Rochester Medical Center, Rochester, New York
  - Albert Einstein Cancer Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Jewish Hospital, The, Cincinnati, Ohio
  - Cleveland Clinic, The, Cleveland, Ohio
  - Mercy Clinic Oncology, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Charles A. Sammons Cancer Center / Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Benaroya Research Institute/Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
- Australia (13):
  - Royal Adelaide Hospital, Adelaide
  - Moorabbin Hospital, Bentleigh East
  - Icon Cancer Care Chermside, Chermside
  - Icon Cancer Care South Brisbane, Chermside
  - Icon Cancer Care Southport, Chermside
  - Icon Cancer Care Wesley, Chermside
  - Monash Medical Centre, Clayton
  - Concord Repatriation General Hospital, Concord
  - St. Vincent's Hospital Sydney, Darlinghurst
  - St Vincent's Public Hospital Sydney - Fitzroy, Fitzroy
  - Western Hospital, Footscray
  - Austin Health, Heidelberg
  - Calvary Mater Newcastle, Waratah
- Canada (4):
  - McGill University Department of Oncology / McGill University Health Centre, Montreal
  - Jewish General Hospital, Montreal
  - Sunnybrook Health Sciences Centre, Toronto
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove-oddeleni klinicke hematologie, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (3):
  - Aarhus University Hospital, Aarhus C
  - Rigs Hospiltalet, Copenhagen
  - Odense University Hospital, Odense C
- France (14):
  - Hôpital Henri Mondor, Créteil
  - CHD Vendée, Site de La Roche-sur-Yon, Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Clinique Victor Hugo, Le Mans
  - CHRU de Lille, Lille
  - Centre Hospitalier Universitaire (CHU) De Limoges - Hopital Dupuytren, Limoges
  - Centre Hospitalier Universitaire Nantes-Hotel Dieu, Nantes
  - Groupe Hospitalier Pitié-Salpétrière, Paris
  - Hopital Saint-Louis / Service d'Hematologie, Paris
  - Groupe Hospitalier du Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rennes, Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel / Centre Regional de Lutte Contre le Cancer, Rouen
- Germany (13):
  - Charite Universitatsmedizin Berlin, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Koln, Cologne
  - Universitatsklinikum Essen, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - Georg-August-Universität Göttingen, Göttingen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinik für Innere Medizin II, Friedrich-Schiller-Universität, Jena
  - Klinikum der Ludwig-Maximilians-Universität München, München
  - Klinikum Nürnberg, Nuremberg
  - Universitätsklinikum Ulm, Ulm
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Israel (5):
  - Soroka Medical Center, Dept. of Oncology, Beersheba
  - Rambam Health Corp., Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (14):
  - Azienda Ospedaliera SS. Antonio E. Biagio E. Cesare Arrigo di Alessandria, Alessandria
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Instituto di Ematologia ed Oncologia Medica, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera-Universitaria Vittorio Emanuele-Ferrarotto-Santo Bambino, Catania
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Niguarda Ca' Granda, Milan
  - IRCSS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Università degli Studi di Roma "La Sapienza, Policlinico Umberto I, Roma
  - Istituto Clinico Humanitas-Humanitas Cancer Center, Rozzano
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Poland (4):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. Ks. B. Markiewicza, Brzozów
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespól Szpitali Miejskich, Chorzów
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Centrum Onkologii Institut im. Marii Sklodowskiej-Curie, Warsaw
- Romania (4):
  - Institutul Clinic Fundeni, Centrul de Hematologie si Transplant Medular Stefan Berceanu, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Institutul Oncologic "Prof. Dr. I. Chiricuta" Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Sectia Clinica Hematologie si Transplant Medular, Târgu Mureş
- South Korea (8):
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (11):
  - Hospital de la Santa Creu i Sant Paul, Barcelona
  - Institut Universitari Dexeus, Barcelona
  - Institut Català D'oncologia, L'Hospitalet de Llobregat
  - Hospital de León, León
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitaro de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (4):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital - Taoyuan, Taoyuan District
- United Kingdom (6):
  - Addenbrooke's Hospital, Cambridge
  - University Hospitals of Leicester NHS Trust, Leicester
  - Saint George's Hospital NHS Trust, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Iyer S, Mehta-Shah N, Advani R, Bartlett NL, Christensen JH, Morschhauser F, Domingo-Domenech E, Rossi G, Kim WS, Alpdogan O, Feldman TA, Camus V, Gritti G, Zinzani PL, Belada D, Mayer J, Choi I, Cheong JW, Rustia E, Fenton K, Fanale M, Savage KJ, Horwitz SM. Association of PET4 response with outcomes of BV-CHP vs CHOP in the ECHELON-2 trial in CD30+ peripheral T-cell lymphoma. Blood Adv. 2025 Dec 9;9(23):5976-5987. doi: 10.1182/bloodadvances.2024015282. PMID 40829107
- [Derived] Domingo-Domenech E, Pro B, Illidge T, Horwitz S, Trumper L, Iyer S, Advani R, Bartlett NL, Christensen JH, Kim WS, Feldman T, Choi I, Gritti G, Belada D, Shustov A, Illes A, Zinzani PL, Huttmann A, Trneny M, Le Gouill S, Jagadeesh D, Friedberg JW, Little M, Dong C, Fanale M, Fenton K, Savage KJ. Brentuximab vedotin plus chemotherapy for the treatment of front-line systemic anaplastic large cell lymphoma: subgroup analysis of the ECHELON-2 study at 5 years' follow-up. Blood Cancer J. 2025 Aug 1;15(1):129. doi: 10.1038/s41408-025-01329-2. PMID 40750774
- [Derived] Savage KJ, Horwitz SM, Advani R, Christensen JH, Domingo-Domenech E, Rossi G, Morschhauser F, Alpdogan O, Suh C, Tobinai K, Shustov A, Trneny M, Yuen S, Zinzani PL, Trumper L, Ilidge T, O'Connor OA, Pro B, Miao H, Bunn V, Fenton K, Fanale M, Puhlmann M, Iyer S. Role of stem cell transplant in CD30+ PTCL following frontline brentuximab vedotin plus CHP or CHOP in ECHELON-2. Blood Adv. 2022 Oct 11;6(19):5550-5555. doi: 10.1182/bloodadvances.2020003971. PMID 35470385
- [Derived] Horwitz S, O'Connor OA, Pro B, Illidge T, Fanale M, Advani R, Bartlett NL, Christensen JH, Morschhauser F, Domingo-Domenech E, Rossi G, Kim WS, Feldman T, Lennard A, Belada D, Illes A, Tobinai K, Tsukasaki K, Yeh SP, Shustov A, Huttmann A, Savage KJ, Yuen S, Iyer S, Zinzani PL, Hua Z, Little M, Rao S, Woolery J, Manley T, Trumper L; ECHELON-2 Study Group. Brentuximab vedotin with chemotherapy for CD30-positive peripheral T-cell lymphoma (ECHELON-2): a global, double-blind, randomised, phase 3 trial. Lancet. 2019 Jan 19;393(10168):229-240. doi: 10.1016/S0140-6736(18)32984-2. Epub 2018 Dec 4. PMID 30522922
- [Derived] Fanale MA, Horwitz SM, Forero-Torres A, Bartlett NL, Advani RH, Pro B, Chen RW, Davies A, Illidge T, Huebner D, Kennedy DA, Shustov AR. Brentuximab vedotin in the front-line treatment of patients with CD30+ peripheral T-cell lymphomas: results of a phase I study. J Clin Oncol. 2014 Oct 1;32(28):3137-43. doi: 10.1200/JCO.2013.54.2456. Epub 2014 Aug 18. PMID 25135998

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Jan2013-Nov2016
Groups:
- A+CHP: brentuximab vedotin, cyclophosphamide, doxorubicin, and prednisone brentuximab vedotin: 1.8 mg/kg every 3 weeks by IV infusion for 6-8 cycles doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for 6-8 cycles prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for 6-8 cycles cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for 6-8 cycles
- CHOP: cyclophosphamide, doxorubicin, vincristine, and prednisone doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for 6-8 cycles prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for 6-8 cycles vincristine: 1.4 mg/m2 (maximum 2 mg) every 3 weeks by IV infusion for 6-8 cycles cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for 6-8 cycles
Period: Overall Study
Arm/Group | A+CHP | CHOP
Started | 226 | 226
Completed (Completed due to study closure by sponsor) | 131 | 116
Not Completed | 95 | 110
Not completed — Withdrawal by Subject | 22 | 16
Not completed — Lost to Follow-up | 3 | 5
Not completed — Death | 68 | 89
Not completed — Not eligible, no study drug received | 1 | 0
Not completed — Change of diagnosis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A+CHP | CHOP | Total
Number analyzed (Participants) | 226 | 226 | 452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 157 | 156 | 313
  >=65 years | 69 | 70 | 139
Age, Continuous [Median (Full Range); unit: years] | 58 [18 to 85] | 58 [18 to 83] | 58 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 75 | 168
  Male | 133 | 151 | 284
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 14
  Not Hispanic or Latino | 186 | 193 | 379
  Unknown or Not Reported | 30 | 29 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45 | 54 | 99
  Black or African American | 12 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 139 | 142 | 281
  Other | 3 | 2 | 5
  Unknown | 26 | 22 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 57 | 127
  Japan | 20 | 23 | 43
  South Korea | 17 | 23 | 40
  Italy | 17 | 20 | 37
  France | 18 | 18 | 36
  Germany | 15 | 12 | 27
  Spain | 15 | 11 | 26
  Czechia | 10 | 12 | 22
  United Kingdom | 7 | 14 | 21
  Australia | 6 | 8 | 14
  Denmark | 9 | 5 | 14
  Israel | 8 | 4 | 12
  Hungary | 4 | 5 | 9
  Taiwan, Province Of China | 5 | 4 | 9
  Poland | 2 | 5 | 7
  Canada | 3 | 3 | 6
  Romania | 0 | 2 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead. One participant (ECOG=0) was assessed after start of treatment.
  Participants
    Grade 0 | 85 | 93 | 178
    Grade 1 | 90 | 86 | 176
    Grade 2 | 51 | 47 | 98

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Per Independent Review Facility (IRF)
Description: The time from the date of randomization to the date of first documentation of progressive disease (PD), death due to any cause, or receipt of subsequent anticancer chemotherapy to treat residual or progressive disease whichever occurred first.
Time Frame: Up to 60 months
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized patients. Patients are included in the treatment group assigned at randomization regardless of the actual treatment received.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | A+CHP | CHOP
Number analyzed (Participants) | 226 | 226
months | 48.20 [8.87 to NA] — Insufficient number of participants experienced events | 20.80 [4.70 to NA] — Insufficient number of participants with events

2. Secondary Outcome: Progression-free Survival Per IRF in Patients With Systemic Anaplastic Large Cell Lymphoma (sALCL)
Description: as for outcome 1
Time Frame: Up to 60 months
Population: This analysis population includes only patients with systemic anaplastic large cell lymphoma (sALCL).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | A+CHP | CHOP
Number analyzed (Participants) | 162 | 154
months | 55.66 [15.61 to NA] — Insufficient number of participants experienced events | 32.03 [4.57 to NA] — Insufficient number of participants experienced events

3. Secondary Outcome: Complete Remission (CR) Rate Per IRF at End of Treatment (EOT)
Description: The count of participants with CR per IRF following the completion of study treatment (at end of treatment or at the first assessment after the last dose of study treatment and prior to long-term follow-up) according to the Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to 8.34 months
Population: The ITT Analysis Set includes all randomized patients. Patients are included in the treatment group assigned at randomization regardless of the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | A+CHP | CHOP
Number analyzed (Participants) | 226 | 226
Participants | 153 | 126

4. Secondary Outcome: Overall Survival (OS)
Description: The time from randomization to death due to any cause.
Time Frame: Up to 90 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | A+CHP | CHOP
Number analyzed (Participants) | 226 | 226
Months | NA [0.0 to 86.5] — The median and 75th percentile of OS was not reached in either treatment arm. The 25th percentile of OS in the A+CHP arm was 40.9 months as compared with 17.5 months in the CHOP arm. | NA [0.1 to 90.0] — The median and 75th percentile of OS was not reached in either treatment arm. The 25th percentile of OS in the A+CHP arm was 40.9 months as compared with 17.5 months in the CHOP arm.

5. Secondary Outcome: Objective Response Rate (ORR) Per IRF at End of Treatment
Description: The count of participants with CR or partial response (PR) per IRF following the completion of study treatment (at end of treatment or the first assessment after the last dose of study treatment and prior to long-term follow-up) according to the Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to 8.34 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | A+CHP | CHOP
Number analyzed (Participants) | 226 | 226
Participants | 188 | 163

6. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Any untoward medical occurrence in a clinical investigational participant administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 8.28 months
Population: The Safety Analysis Set includes all patients who receive any amount of brentuximab vedotin or any component of CHOP. Treatment group will be determined using the actual treatment received, regardless of the randomization treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | A+CHP | CHOP
Number analyzed (Participants) | 223 | 226
Participants
  Any treatment-emergent AE | 221 | 221
  Blinded study treatment-related AE | 201 | 193
  CHP treatment-related AE | 198 | 205
  Any serious adverse event (SAE) | 87 | 87
  Blinded study treatment-related SAE | 58 | 45
  CHP treatment-related SAE | 62 | 53
  Treatment discontinuations due to AE | 14 | 15
  Treatment discontinuations due to blinded study treatment-related AE | 10 | 10
  Treatment discontinuations due to CHP treatment-related AE | 8 | 7

7. Secondary Outcome: Incidence of Laboratory Abnormalities
Description: Number of participants who experienced a Grade 3 or higher laboratory toxicity.
Time Frame: Up to 8.28 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | A+CHP | CHOP
Number analyzed (Participants) | 223 | 226
Participants
  Any Chemistry Test | 25 | 23
  Alanine Aminotransferase High | 3 | 1
  Albumin Low | 2 | 3
  Alkaline Phosphatase High | 1 | 0
  Calcium Low | 1 | 1
  Glucose High | 8 | 6
  Phosphate Low | 4 | 3
  Potassium High | 0 | 2
  Potassium Low | 3 | 2
  Sodium High | 1 | 0
  Sodium Low | 4 | 6
  Urate High | 5 | 2
  Any Hematology Test | 68 | 78
  Absolute Neutrophil Count Low | 17 | 19
  Hemoglobin High | 1 | 0
  Hemoglobin Low | 9 | 13
  Leukocytes Low | 12 | 21
  Lymphocytes High | 0 | 1
  Lymphocytes Low | 52 | 61
  Neutrophils Low | 17 | 19
  Platelets Low | 1 | 1

ADVERSE EVENTS:
Time Frame: Non-serious AEs followed up to 8 months. Serious AEs followed up to 90 months
Description: Safety Analysis Population: Includes all randomized participants who received at least one dose of study treatment.
  Investigator and study personnel report all adverse events (AEs) and serious adverse events (SAEs) whether elicited during patient questioning, discovered during physical examination, laboratory testing and/or other means.
Groups:
- A+CHP Subgroup: Includes only participants in A+CHP arm who were randomized but did not receive treatment.
Arm/Group | A+CHP | CHOP | A+CHP Subgroup
All-Cause Mortality (participants affected / at risk) | 67/223 | 89/226 | 1/3
Serious Adverse Events (participants affected / at risk) | 89/223 | 90/226 | 0/0
Other Adverse Events (participants affected / at risk) | 220/223 | 218/226 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A+CHP (N=223) | CHOP (N=226) | A+CHP Subgroup (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 32 | 26 | 0
Pneumonia (Infections and infestations) | 11 | 3 | 0
Pyrexia (General disorders) | 9 | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 6 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Sepsis (Infections and infestations) | 5 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 0
Device related infection (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Neutropenic infection (Infections and infestations) | 2 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abscess soft tissue (Infections and infestations) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Anal fistula infection (Infections and infestations) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0
Extravasation (General disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Infection (Infections and infestations) | 1 | 1 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0
Injection site infection (Infections and infestations) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Septic shock (Infections and infestations) | 1 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 11 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
CSF volume decreased (Investigations) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Device issue (Product Issues) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 3 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Ulcerative gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A+CHP (N=223) | CHOP (N=226) | A+CHP Subgroup (N=0)
Neutropenia (Blood and lymphatic system disorders) | 87 | 81 | NA
Anaemia (Blood and lymphatic system disorders) | 64 | 49 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 14 | NA
Leukopenia (Blood and lymphatic system disorders) | 18 | 13 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 9 | NA
Hypothyroidism (Endocrine disorders) | 12 | 11 | NA
Nausea (Gastrointestinal disorders) | 114 | 91 | NA
Constipation (Gastrointestinal disorders) | 98 | 94 | NA
Diarrhoea (Gastrointestinal disorders) | 93 | 55 | NA
Vomiting (Gastrointestinal disorders) | 60 | 37 | NA
Stomatitis (Gastrointestinal disorders) | 28 | 27 | NA
Abdominal pain (Gastrointestinal disorders) | 26 | 22 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22 | 16 | NA
Abdominal pain upper (Gastrointestinal disorders) | 23 | 10 | NA
Dyspepsia (Gastrointestinal disorders) | 17 | 12 | NA
Haemorrhoids (Gastrointestinal disorders) | 8 | 12 | NA
Fatigue (General disorders) | 83 | 80 | NA
Pyrexia (General disorders) | 86 | 74 | NA
Oedema peripheral (General disorders) | 40 | 36 | NA
Asthenia (General disorders) | 35 | 20 | NA
Mucosal inflammation (General disorders) | 15 | 14 | NA
Chest pain (General disorders) | 14 | 8 | NA
Malaise (General disorders) | 8 | 12 | NA
Upper respiratory tract infection (Infections and infestations) | 18 | 12 | NA
Nasopharyngitis (Infections and infestations) | 10 | 12 | NA
Urinary tract infection (Infections and infestations) | 12 | 9 | NA
Weight decreased (Investigations) | 54 | 43 | NA
Alanine aminotransferase increased (Investigations) | 11 | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 53 | 47 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 24 | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 14 | 13 | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 12 | NA
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 | 13 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 9 | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 9 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 43 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 20 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 21 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 21 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 12 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 112 | 108 | NA
Headache (Nervous system disorders) | 37 | 36 | NA
Dizziness (Nervous system disorders) | 32 | 24 | NA
Paraesthesia (Nervous system disorders) | 13 | 19 | NA
Dysgeusia (Nervous system disorders) | 13 | 15 | NA
Peripheral motor neuropathy (Nervous system disorders) | 8 | 18 | NA
Insomnia (Psychiatric disorders) | 52 | 49 | NA
Anxiety (Psychiatric disorders) | 30 | 13 | NA
Depression (Psychiatric disorders) | 16 | 15 | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 9 | 14 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 44 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 33 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 19 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 58 | 56 | NA
Night sweats (Skin and subcutaneous tissue disorders) | 46 | 63 | NA
Rash (Skin and subcutaneous tissue disorders) | 27 | 21 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 15 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 17 | NA
Hypertension (Vascular disorders) | 71 | 68 | NA
Hypotension (Vascular disorders) | 15 | 14 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT01777152/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT01777152/SAP_001.pdf